CLINICAL TRIAL: NCT06641115
Title: Integrated Treatment for Co-Occurring Opioid Use Disorder and Posttraumatic Stress Disorder
Brief Title: Integrated Treatment for Opioid Use Disorder and PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00138487; K23DA055209 (NIH)
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder; Posttraumatic Stress Disorder (PTSD)
Keywords: Mental Health; Psychiatry; Substance Use; PTSD; Opioid Use; Therapy
MeSH Terms: conditions — Opioid-Related Disorders; Stress Disorders, Post-Traumatic; Psychological Well-Being; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOPE Therapy (Experimental): Helping Opioid Use and PTSD with Exposure (HOPE) therapy is an integrated 10-12 week treatment for opioid use disorder and trauma/posttraumatic stress disorder
  Interventions: Behavioral: HOPE Therapy
- Treatment as Usual (No Intervention): Participants take medications as prescribed and attend standard community substance use treatment services

INTERVENTIONS:
Behavioral: HOPE Therapy — Helping Opioid Use and PTSD with Exposure (HOPE) therapy is an integrated 10-12 week treatment for opioid use disorder and trauma/posttraumatic stress disorder
  Arms: HOPE Therapy

SUMMARY:
This study will test a therapy intervention, HOPE, for individuals with opioid use disorder and posttraumatic stress disorder. Interested individuals will need to be taking medications for opioid use disorder (e.g., suboxone, naltrexone, methadone). Interested participants will complete a 10-12 week therapy, and be asked to complete surveys.

DETAILED DESCRIPTION:
Up to half of individuals with OUD have PTSD, but to date, there are no established evidence-based behavioral interventions that concurrently address OUD and PTSD symptoms. The proposed study directly addresses this major clinical gap by testing whether augmenting medications for OUD by testing an adapted, trauma-focused, integrated behavioral treatment for substance use disorders and co-occurring PTSD (i.e., Helping Opioid Use and PTSD with Exposure; HOPE) will enhance clinical outcomes. The investigators will test HOPE combined with medications for OUD (MOUD) versus MOUD-only in a randomized clinical trial among 76 individuals with OUD and PTSD to evaluate feasibility and preliminary efficacy in reducing opioid use and PTSD severity. Both conditions will also complete ecological momentary assessments (EMA) to assess for daily opioid use, craving, and PTSD symptoms. EMA will allow for the assessment of the associations between daily PTSD symptoms and opioid craving and use, which may then inform treatment development.

ELIGIBILITY:
Inclusion Criteria:

* Any gender; any race or ethnicity; aged 18-70 years old.
* English-speaking
* Meet DSM-5 diagnostic criteria for OUD.
* Meet DSM-5 diagnostic criteria for PTSD and have some memory of their index traumatic event.
* Must be maintained on a stable dose of medication for OUD for at least 1 month.
* Participants taking psychotropic medications will be required to be maintained on a stable dose for at least 1 month before study initiation.

Exclusion Criteria:

* Participants presenting with psychiatric contraindications (e.g., unmanaged psychosis or mania, or bipolar) will be excluded and referred clinically.
* Participants considered an immediate suicide risk, with current suicidal ideation and a plan of intent, or displaying other high-risk behaviors (i.e., MOUD refusal, risky fentanyl use, etc.), as determined by the PI and study team. These individuals will complete a safety plan and be referred for treatment.
* Participants meeting DSM-5 criteria for a concurrent, non-opioid, substance use disorder and who report that the other substance is their primary substance of use. These participants will be referred clinically for treatment.
* Participants enrolled in ongoing evidence-based psychotherapy for substance use disorders or PTSD outside of medications for OUD and standard psychotherapy groups in treatment programs.
* Medical problems requiring immediate and intensive treatment, such as unstable or symptomatic end stage liver disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Opioid Use | through study treatment completion, an average of 12 weeks
  Opioid use (percent days using) as measured by urine drug screens
Change in Posttraumatic Stress Disorder Symptoms | through study treatment completion, an average of 12 weeks
  Posttraumatic Stress Disorder symptoms as measured by the Clinician Administered Posttraumatic Stress Disorder Scale for the Diagnostic and Statistical Manual for Mental Disorders, 5th Edition or the CAPS-5. Total severity scores on this measure range from 0-80 with higher scores denoting more severe posttraumatic stress disorder symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Saraiya, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No